CLINICAL TRIAL: NCT01886742
Title: Adequacy of Perioperative Cefazolin for Surgery Antibiotic Prophylaxis in Obese Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1653
Record Dates: First submitted 2013-02-28; First posted 2013-06-26 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Obesity
Keywords: Perioperative antibiotic prophylaxis; Morbidly Obese
MeSH Terms: conditions — Obesity | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard dose group (2 g intravenous (IV) cefazolin dose for patients <120 kg, and 3 g IV cefazolin for patients >120 kg)
  Interventions: Drug: Standard Dose Group
- Treatment group (Experimental): Weight-based dose group (30 mg/kg cefazolin IV)
  Interventions: Drug: Weight Based Group

INTERVENTIONS:
Drug: Standard Dose Group — The standard dose of Cefazolin will be administered intravenously.
  Arms: Control group
Drug: Weight Based Group — The weight-based dose group will receive 30 mg/kg cefazolin dose intravenously.
  Arms: Treatment group

SUMMARY:
The population continues to increase in weight. Currently there are no guidelines in the dosing of cefazolin for the obese population. Standard dosing of cefazolin 2 grams for patients <120 kg and 3 grams for patients >120 kg is used as the dose for surgical prophylaxis. This makes no provisions for weight based dosing. There has been some recent data which states this might not be enough for the obese patients. The primary objective of this study is to determine if weight based dosing (30 mg/kg) of cefazolin as surgical prophylaxis for patients undergoing elective gastric bypass/laparoscopic Roux-en-y gastric bypass provides appropriate serum concentrations for a larger percentage of time than the current method of giving the standard 2 or 3 gram doses of cefazolin peri-operatively. The concentration of cefazolin in tissue will also be measured to help assess this question.

DETAILED DESCRIPTION:
The hypothesis of this study is that customary doses of antibiotics, when administered for perioperative surgical prophylaxis, are insufficient to achieve adequate antibiotic concentrations in blood and tissues of morbidly obese patients (defined as a BMI greater than 40 kg/m2) and that these patients are therefore placed at high risk of surgical wound infections and poor clinical outcomes. Cefazolin is a first-generation cephalosporin commonly used for perioperative surgical prophylaxis in colorectal, abdominal, bariatric, gynecologic and obstetric, or orthopedic total joint arthroplasty surgical procedures. Previous cefazolin pharmacokinetic (PK) analysis in obese patients led to conflicting results and recommendations. It is not clearly know to what extent the pharmacokinetics of cefazolin in morbidly obese patients differ from those of non-obese patients. Specific dosing guidelines are then lacking. The main objective of this study is to assess the pharmacokinetics of cefazolin in morbidly obese after administrations of a standard recommended 2-3 g dose or a weight-base 30-mg/kg dose

ELIGIBILITY:
Inclusion Criteria:

1. BMI greater than 40
2. No known history of allergy to cephalosporins
3. Scheduled for elective gastric bypass or laparoscopic Roux-en-y gastric bypass procedures
4. Able to read and understand English

Exclusion Criteria:

1. Patients <18 years of age or >89 Years of age
2. Pregnant women, prisoners and decisionally challenged subjects will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Pharmacokinetics of Cefazolin in the Morbidly Obese | Before cefazolin admin., then at 10, 30, 60, 120, 180 minutes after injection and at wound closure.
  Since the goal of perioperative antimicrobial prophylaxis is to achieve free (unbound) serum and tissue drug levels that exceed the MIC for likely pathogens across the duration of the surgical procedure, and since redosing of cefazolin is recommended every 3-4 hours, PK/PD performance of cefazolin over that time frame will be analyzed. For the purposes of this study, pharmacodynamic targets are defined as fT>MIC (time during which free drug concentrations exceed pathogen MICs) of 100% over periods of up to 4 hours in duration. The PK/PD probability of target attainment (PTA) for pharmacodynamic goals and the cumulative fraction of response (CFR) for both cefazolin regimens will be compared. A PTA of ≥90% and a CFR of ≥ 90% for a dosage regimen (i.e., predicted to meet pharmacodynamic targets in ≥ 90% of the total bacterial population across the full range of MICs) are considered optimum.

SECONDARY OUTCOMES:
Incidence of surgical site infection | Within 1 month postoperatively
  The incidence of surgical site infection will be monitored and compared.
Hospital length of stay | Hospital discharge
  The length of time the subject is hospitalized will be monitored and compared.
Hospital readmission | Witihn 1 month after hospital discharge
  Hospital readmission within 1 month postoperatively.
Incidence of adverse outcomes | Within 1 month postoperatively
  Adverse outcomes in these patients will be monitored and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Moine, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No